CLINICAL TRIAL: NCT04578860
Title: A 3-months, Controlled and Double-blind Trial of the Effectiveness of Music Therapy in the Treatment of Sleep Disorders in General Medicine.
Brief Title: Effectiveness of Music Therapy on Sleep Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Saint-Quentin-en-Yvelines University (Other)
Responsible Party: Principal Investigator, MUSSO, PhD student in medicine, Versailles Saint-Quentin-en-Yvelines University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19.05.07.57052
Record Dates: First submitted 2020-09-03; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Sleep Disorder; Chronic Insomnia
Keywords: music therapy; white noise; sleeping medicine; psychotropics
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (Active Comparator): Usual treatment of sleep disorders consist of adequate sleep hygiene entails the behaviors, practices, rituals, and habits.
  Interventions: Other: Treatment as usual for sleep disorders
- Music Intervention (Experimental): Using the app Music Care
  Interventions: Other: Music therapy with Music Care app
- White Noise (Placebo Comparator): Using an app producing white noise (like rain, storm, fan, wind...)
  Interventions: Other: Sound therapy with White Noise

INTERVENTIONS:
Other: Music therapy with Music Care app — Listening to music with Music Care app, every day, for 20 minutes, sitting up or lying down, at bedtime, with a headset or earbuds.
  Arms: Music Intervention
Other: Sound therapy with White Noise — Listening to white noise with an app, every day, for 20 minutes, sitting up or lying down, at bedtime, with a headset or earbuds.
  Arms: White Noise
Other: Treatment as usual for sleep disorders — No intervention
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to determine whether listening to music before falling asleep can improve sleep quality in patients with sleep disorders.

DETAILED DESCRIPTION:
Sleep is a key factor in a person's health, and we actually spend one third of our lives sleeping. The latest figures show a prevalence of insomnia in 20-30% of French adults. Sleep disorders are a growing public health concern.

Treatment for insomnia is often some form of drugs; however, the side effects of these treatments (sedatives, hypnotics or anti-anxiety medications) are significant. Non drug-treatments like music therapy are growing in popularity. The objective of this study is to demonstrate the effectiveness of musical interventions on sleep disorders in general population.

It is a prospective, multicentered, double-blind, randomized comparative intervention study, comparing 3 parallel patient groups. Patients included in this study will be selected by their physicians according to the severity of their disorders. Enrollment period will last for 2 months and the study will last 3 months. The primary outcome (score on Pittsburgh Sleep Quality Index, PSQI) is a discrete quantitative variable. The statistical tests used will concern the comparison of the average deltas of each group by using analysis of variance (ANOVA). The selected alpha risk, or Type 1 error, is 5%.

The results expected in this study are a significant decrease in Pittsburgh scale scores in the music intervention group. The decrease in Pittsburgh scale scores should be compared to the results from this study: Qun Wang and Al; The Effects of Music Intervention on Sleep Quality in Community-Dwelling Elderly, The Journal of Alternative and Complementary Medicine, 2016. In this 3-month study, the average change compared to the baseline is 6.44 in the musical intervention group and 3.28 in the control group. The pooled standard deviation is estimated to be 3.53.

Musical intervention is non-invasive, so it's a low-risk therapeutic tool for general practice that may be useful in the management of sleep disorders. Its effectiveness, if demonstrated, could lead to new recommendations for the treatment of sleep disorders, and reduce the use of medication such as sedatives and hypnotics.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years old
* speaking French,
* with sleep complaints at least 3 times a week for more than 3 months,
* or with a sleep medications at least 3 times a week for more than 3 months,
* and an ISI score (Insomnia Severity Index) greater than 14

Exclusion Criteria:

* Age < 18 years old.
* Patients with severe cognitive disorders or comprehension disorders deemed incompatible with the study protocol by the physician.
* Patients with severe hearing loss, not using hearing aids.
* Patients who do not own a music distribution device (smartphone, tablet, laptop, hifi system...).
* Patients without internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Score on Pittsburgh Sleep Quality Index (PSQI) | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.

SECONDARY OUTCOMES:
Severity of anxiety | 3 months
  Evaluate the effect of musical interventions and white noise on patient anxiety at the beginning, during, and at the end of the study (in a scale between 1 and 4).
Quantity of sleeping medications used per week | 3 months
  Evaluate the effect of musical interventions and white noise on the quantity of sleeping medications used per week for sleeping at the beginning and end of the study.
Patient's overall state of well-being | 3 months
  Evaluation of the patient's overall state of well-being with one simple question: How do you find your health status now as compared to the beginning of the study? (Worse/No change/Slight change/Noticeable change).

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Musso, Principal Investigator — Versailles Saint-Quentin-en-Yvelines University
Locations (1):
- Versailles-Saint Quentin en Yvelines University, Versailles, Île-de-France Region, France

REFERENCES:
- [Background] Harmat L, Takacs J, Bodizs R. Music improves sleep quality in students. J Adv Nurs. 2008 May;62(3):327-35. doi: 10.1111/j.1365-2648.2008.04602.x. PMID 18426457
- [Background] Jespersen KV, Koenig J, Jennum P, Vuust P. Music for insomnia in adults. Cochrane Database Syst Rev. 2015 Aug 13;2015(8):CD010459. doi: 10.1002/14651858.CD010459.pub2. PMID 26270746
- [Background] Blais FC, Gendron L, Mimeault V, Morin CM. [Evaluation of insomnia: validity of 3 questionnaires]. Encephale. 1997 Nov-Dec;23(6):447-53. French. PMID 9488928
- [Result] Gottlieb DJ, Redline S, Nieto FJ, Baldwin CM, Newman AB, Resnick HE, Punjabi NM. Association of usual sleep duration with hypertension: the Sleep Heart Health Study. Sleep. 2006 Aug;29(8):1009-14. doi: 10.1093/sleep/29.8.1009. PMID 16944668
- [Result] Gangwisch JE, Heymsfield SB, Boden-Albala B, Buijs RM, Kreier F, Pickering TG, Rundle AG, Zammit GK, Malaspina D. Short sleep duration as a risk factor for hypertension: analyses of the first National Health and Nutrition Examination Survey. Hypertension. 2006 May;47(5):833-9. doi: 10.1161/01.HYP.0000217362.34748.e0. Epub 2006 Apr 3. PMID 16585410
- [Result] Spiegel K, Knutson K, Leproult R, Tasali E, Van Cauter E. Sleep loss: a novel risk factor for insulin resistance and Type 2 diabetes. J Appl Physiol (1985). 2005 Nov;99(5):2008-19. doi: 10.1152/japplphysiol.00660.2005. PMID 16227462
- [Result] Leger D, Guilleminault C, Dreyfus JP, Delahaye C, Paillard M. Prevalence of insomnia in a survey of 12,778 adults in France. J Sleep Res. 2000 Mar;9(1):35-42. doi: 10.1046/j.1365-2869.2000.00178.x. PMID 10733687
- [Result] Young TB. Epidemiology of daytime sleepiness: definitions, symptomatology, and prevalence. J Clin Psychiatry. 2004;65 Suppl 16:12-6. PMID 15575799
- [Result] Feng F, Zhang Y, Hou J, Cai J, Jiang Q, Li X, Zhao Q, Li BA. Can music improve sleep quality in adults with primary insomnia? A systematic review and network meta-analysis. Int J Nurs Stud. 2018 Jan;77:189-196. doi: 10.1016/j.ijnurstu.2017.10.011. Epub 2017 Oct 23. PMID 29100201
- [Result] Wang CF, Sun YL, Zang HX. Music therapy improves sleep quality in acute and chronic sleep disorders: a meta-analysis of 10 randomized studies. Int J Nurs Stud. 2014 Jan;51(1):51-62. doi: 10.1016/j.ijnurstu.2013.03.008. Epub 2013 Apr 9. PMID 23582682
- [Result] Guetin S, Coudeyre E, Picot MC, Ginies P, Graber-Duvernay B, Ratsimba D, Vanbiervliet W, Blayac JP, Herisson C. [Effect of music therapy among hospitalized patients with chronic low back pain: a controlled, randomized trial]. Ann Readapt Med Phys. 2005 Jun;48(5):217-24. doi: 10.1016/j.annrmp.2005.02.003. Epub 2005 Mar 4. French. PMID 15914256
- [Result] Guetin S, Portet F, Picot MC, Pommie C, Messaoudi M, Djabelkir L, Olsen AL, Cano MM, Lecourt E, Touchon J. Effect of music therapy on anxiety and depression in patients with Alzheimer's type dementia: randomised, controlled study. Dement Geriatr Cogn Disord. 2009;28(1):36-46. doi: 10.1159/000229024. Epub 2009 Jul 23. PMID 19628939
- [Result] Jaber S, Bahloul H, Guetin S, Chanques G, Sebbane M, Eledjam JJ. [Effects of music therapy in intensive care unit without sedation in weaning patients versus non-ventilated patients]. Ann Fr Anesth Reanim. 2007 Jan;26(1):30-8. doi: 10.1016/j.annfar.2006.09.002. Epub 2006 Nov 3. French. PMID 17085009
- [Result] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Result] Guetin S, Portet F, Picot MC, Defez C, Pose C, Blayac JP, Touchon J. [Impact of music therapy on anxiety and depression for patients with Alzheimer's disease and on the burden felt by the main caregiver (feasibility study)]. Encephale. 2009 Feb;35(1):57-65. doi: 10.1016/j.encep.2007.10.009. Epub 2008 Feb 20. French. PMID 19250995
- [Result] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Result] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Result] Savard MH, Savard J, Simard S, Ivers H. Empirical validation of the Insomnia Severity Index in cancer patients. Psychooncology. 2005 Jun;14(6):429-41. doi: 10.1002/pon.860. PMID 15376284
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Edinger JD, Wohlgemuth WK. Psychometric comparisons of the standard and abbreviated DBAS-10 versions of the dysfunctional beliefs and attitudes about sleep questionnaire. Sleep Med. 2001 Nov;2(6):493-500. doi: 10.1016/s1389-9457(01)00078-8. PMID 14592264
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Result] Wang Q, Chair SY, Wong EM, Li X. The Effects of Music Intervention on Sleep Quality in Community-Dwelling Elderly. J Altern Complement Med. 2016 Jul;22(7):576-84. doi: 10.1089/acm.2015.0304. Epub 2016 May 25. PMID 27223689
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763
- See also: Centre International de Musicothérapie. Historique du C.I.M — http://musicotherapie.info/le-centre/le-cim/
- See also: Giordanella JP. Rapport sur le thème du sommeil. Ministère de la Santé et des Solidarités. Décembre 2006 — https://solidarites-sante.gouv.fr/IMG/pdf/rapport-5.pdf
- See also: Association Française de Musicothérapie. L'A.F.M et la musicothérapie — https://www.afm-musicotherapie.org/
- See also: Fédération Française de Musicothérapie. Fédération Française de Musicothérapie — https://www.musicotherapie-federationfrancaise.com/missions/